CLINICAL TRIAL: NCT03633409
Title: Differential EBI2 Expression Upon Allelic Status of the rs9557195 Polymorphism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EBI2-Study
Record Dates: First submitted 2018-07-02; First posted 2018-08-16 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; EBI2; G protein coupled receptor; FACS; UBAC2; lymphocyte migration; single nucleotide polymorphism
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD patients and healthy volunteers: We will recruit IBD patients and healthy volunteers

SUMMARY:
EBI2 is a risk gene for inflammatory bowel diseases (rs9557195). Patients of the Swiss IBD cohort study have been genotyped for the allelic status of EBI2. The investigators will test the influence of rs9557195 genoty (TT or CC allel), inflammatory activity and current treatment (infliximab vs. vedolizumab) on expression and activity of EBI2 on blood lymphocytes, mRNA expression of EBI2 and UBAC2 (located on the opposite DNA strand of EBI2) and activity of lymphocytes on a migraton assay.

DETAILED DESCRIPTION:
EBI2 is a risk gene for inflammatory bowel diseases (rs9557195). EBI2 is a G protein coupled receptors expressed on the immune cells. EBI2 directs migration and activity of immune cells.

Patients of the Swiss IBD cohort study have been genotyped for the allelic status of EBI2. The investigators will recruit patients with Crohn's disease and ulcerative colitis, assess epidemiological and clinical parameters (including clinical activity of IBD) draw blood, isolate lymphocytes, DNA and RNA.

The investigators will test the influence of rs9557195 genotype (TT or CC allel), inflammatory activity and current treatment (infliximab vs. vedolizumab) on expression and activity of EBI2 on blood lymphocytes (by FACS using an EBI2-antibody), mRNA expression (by qPCR) of EBI2 and UBAC2 (located on the opposite DNA strand of EBI2) and activity of lymphocytes on a migration assay.

ELIGIBILITY:
Inclusion Criteria:

* Patient with IBD OR healthy volunteer
* No major uncontrolled medical/ surgical/ psychiatric condition requiring ongoing management besides IBD in the respective study groups. Well controlled conditions (i.e. medically controlled arterial hypertension, occupational asthma) may be present

Exclusion Criteria: none

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: we will recruit a mixed population (patients can be in more than one group)
  * up to 100 healthy volunteers
  * up to 30 IBD patients with the rs9557195-CC IBD risk genotype in clinical remission
  * up to 30 IBD patients with the rs9557195-CT IBD risk genotype in clinical remission
  * up to 30 IBD patients with the rs9557195-TT IBD low risk genotype in clinical remission
  * up to 50 IBD patients of any genotype during a flare
  * up to 50 IBD patients of any genotype treated with vedolizumab
  * up to 50 IBD patients of any genotype treated with a TNF-inhibitor (infliximab, adalimumab, golimumab, certolizumab)
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
EBI2 expression - dependent on rs9557195 allele status (FACS) | at time of inclusion into the study
  EBI2 levels in PBMCs will be determined by FACS, and compared according to allele status of rs9557195

SECONDARY OUTCOMES:
EBI2 expression - dependent on rs9557195 allele status (RT-PCR) | at time of inclusion into the study
  EBI2 levels in PBMCs will be determined by RT-PCR, and compared according to EBI2 levels in PBMCs will be determined by RT-PCR, and compared according to allele status of rs9557195
UBAC2 expression - dependent on rs9557195 allele status (RT-PCR) | at time of inclusion into the study
  UBAC2 levels in PBMCs will be determined by RT-PCR, and compared according to 2 levels in PBMCs will be determined by RT-PCR, and compared according to allele status of rs9557195
Motility of PBMCs dependent on rs9557195 allele status (Boyden chamber) | at time of inclusion into the study
  motility of PBMCs will be assessed using the Boyden chamber and compared according to allele status of rs9557195
EBI2-expression (FACS) in individuals treated with infliximab vs. vedolizumab | at time of inclusion into the study
  We will compare EBI2 expression as determined by FACS in individuals with infliximab and vedolizumab treatment
EBI2-expression (FACS) according to gut inflammation | at time of inclusion into the study
  We will compare EBI2 expression (determined by FACS) in IBD patients with severe disease, in remission and in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
some of the outcome measures (EBI2 expression, cell motility assays) will be performed by external collaborators